CLINICAL TRIAL: NCT05093543
Title: Feasibility and Effect of a Multidisciplinary Telematics Approach for Chronic Non-specific Low Back Pain: a Randomized, Open-label, Controlled, Pilot Clinical Trial. Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Iago Garreta Catala, Consultant of Orthopaedics Surgery, Principal Investigator, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUB-COT-ENFORMA-2021
Record Dates: First submitted 2021-05-05; First posted 2021-10-26 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The experimental group is based on a telematic multidisciplinary approach for CnsLBP. Scheduled and periodic telematic sessions will be performed. The multidisciplinary approach (to be carried out by telematic means) consists of a biopsychosocial rehabilitation program for patients with CnsLBP that includes physical rehabilitation/physiotherapy and psychosocial group sessions (performed by psychologists, social workers), which will be offered as part of the integrated program.
  Patients assigned to the experimental group will receive a Google Meet® link by email, so that they may join the weekly 2-hour group sessions (every Tuesday at 9 a.m.). Google Meet® is a free real-time meeting app by Google that does not require download, has no session time limit, and neither limits the number of users per session. Patients assigned to the experimental group will receive a single-use link by email to access each online group session.
  Interventions: Behavioral: physical rehabilitation/physiotherapy and psychosocial group sessions
- Control (No Intervention): Explanation for choice of comparators {6b} The telematics multidisciplinary approach (experimental group) will be compared to Standard of Care (SoC) (control group). SoC consists of a patient's follow up according to the usual clinical practice. In Bellvitge University Hospital's setting, the treatment protocol for CnsLBP indicates physical rehabilitation/physiotherapy as the first treatment step, and Pain Clinic evaluation as a second step for those who did not improve. For patients who did not improve with the previous steps and that still demand a solution for their CnsLBP, a third step would be to refer the patient for surgical evaluation - a spine surgeon would, then, evaluate, alongside with the patient, whether a surgical approach would be appropriate for his/her case. If the surgery is ruled out by the spine surgeon, the patient may be referred, once more, to physical rehabilitation/physiotherapy and/or to the Pain Clinic, at the surgeon's discretion.

INTERVENTIONS:
Behavioral: physical rehabilitation/physiotherapy and psychosocial group sessions — physical rehabilitation/physiotherapy and psychosocial group sessions
  Arms: Intervention

SUMMARY:
Low back pain is a challenging condition, with a lifetime prevalence of up to 84%. The estimated prevalence of chronic non-specific low back pain is of approximately 23%. Although pain is a sensory experience triggered by a peripheral stimulus, psychosocial factors influence on its perception and on the risk of chronification.

Chronic Low Back Pain imposes a substantial socioeconomic burden to patients, families, and healthcare systems worldwide. It is a multifactorial condition, characterized by a combination of physical, psychosocial and occupational factors. We have planned two working hypotheses: (1) coordinating several healthcare professionals is feasible to manage chronic non-specific low back pain through telematics multidisciplinary approach; (2) telematics multidisciplinary approach improves the quality of life of patients with chronic non-specific low back pain and in whom conservative treatment has failed. Hence, we aim to assess the feasibility and effect of telematics multidisciplinary approach in patients suffering from chronic non-specific low back pain and who have not improved with conservative treatment.

Patients will be randomized to the telematics multidisciplinary approach (Experimental Group) or to the Standard of Care (Control Group). Scheduled and periodic telematics multidisciplinary sessions will be performed. Each session will consist of an integrated program that combines rehabilitation (i.e., group-based exercise program), psychological treatment and social work sessions. Standard of Care, after conservative treatment failure, depends mainly on the physician in charge's discretion and on the patients' preferences. An exploratory analysis will be performed.

The results of this clinical trial will provide evidence that a scheduled telematics multidisciplinary approach will improve the quality of life of these patients and empower them to be more autonomous. Likewise, telematics multidisciplinary approach is feasible to manage chronic non-specific low back pain in patients unresponsive to conservative treatment. Consequently, these patients are less likely to wander through different medical specialties seeking for a solution to their condition, presumably avoiding ineffective back surgeries. The results will also highlight the importance of patients playing an active role in their own treatment to successfully manage chronic non-specific low back pain.

DETAILED DESCRIPTION:
Objectives {#7}:

Hypothesis:

Two working hypothesis have been planned: i) the coordination of several health care professionals is feasible to manage CnsLBP (Chronic non-specific Low Back Pain) through telematics multidisciplinary approach; ii) telematics multidisciplinary approach improves the quality of life of patients who suffer from CnsLBP and in whom conservative treatment has failed

Primary Objective The primary aims are to assess the feasibility and effect of the telematics multidisciplinary approach in patients who suffer from non-specific CnsLBP and in whom conservative treatment has failed.

Secondary objectives

The secondary objectives are:

1. to quantify the desertion rate
2. to study the level of usual physical activity
3. to quantify disability due to CnsLBP
4. to study anxiety and depression
5. to assess chronic pain coping strategies
6. to study self-awareness and emotional self-regulation
7. to evaluate perceived social support
8. to estimate mental well-being

Trial Design {#8}:

This is an open-label, randomized, controlled, parallel-group, pilot clinical trial. Patients will be randomized to the telematic multidisciplinary biopsychosocial approach (Experimental Group) or to the Standard of Care (Control Group).

This pilot clinical trial will provide evidence on the feasibility of the coordination of several health care professionals to manage CnsLBP through telematics multidisciplinary approach; and it will provide the first evidence on the impact of the telematics multidisciplinary approach on the QoL of these patients.

The target population will be patients with CnsLBP who have already undergone rehabilitation and pain clinic therapy and are still in pain and seeking for a solution (i.e., patients on a waiting list to see a spine surgeon for surgical assessment, patients who might be candidates to lumbar surgery depending on their evolution, patients being followed up by a Pain Clinic specialist or by their assigned General Practitioner specialist). If during the trial it is decided to perform a lumbar surgical intervention on an included patient, he/she will be automatically excluded from the trial.

Methods: Participants, Interventions and Outcomes

Study Setting {#9}:

This trial will be carried out in the premises of the Bellvitge University Hospital (a tertiary hospital), the Viladecans Hospital (a secondary hospital) and primary care centers: Delta del Llobregat Primary Care Center, L'Hospitalet de Llobregat Mental Health Unit, Santa Eulalia Primary Care Center.

ELIGIBILITY:
Eligibility Criteria {#10}:

Inclusion Criteria:

* Patients between 18 and 67 years of age (i.e., working age population).
* Both genders.
* Patients with chronic non-specific low back pain that does not improve with conservative treatment (including rehabilitation and Pain Clinic evaluation and follow-up).
* The predominant symptom must be low back pain (and not pain radiating to the extremities).
* Patients who sign the informed consent form

Exclusion Criteria:

* Patients who have previously undergone lumbar arthrodesis.
* Patients diagnosed with lumbar instability or non-degenerative pathologies (fractures, tumors, infections, etc.) that justify their chronic low back pain.
* Patients who cannot move independently.
* Patients who have a contraindication to perform light aerobic exercise or physical therapy exercises for the treatment of low back pain.
* Patients with a psychiatric history that interferes with their daily life
* Patients who are possible candidates for low back surgery, with a planned intervention during the study period.
* Patients who have a programmed Pain Clinic intervention or extra rehabilitation sessions scheduled during the study period.
* Patients who lack motivation or show no commitment to the program.
* Patients who do not have access to a device with internet connection and/or to a webcam (smartphone, tablet, or computer).

Note: Since this is a pilot clinical trial with a small sample size, patients who receive extra sessions of rehabilitation or interventions in Pain Clinic will be withdrawn from the study to minimize the impact on the results, although these treatments are also part of the SoC.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Number of sessions performed out of the 8 sessions scheduled | 6 months
  number of telematics multidisciplinary sessions performed out of the 8 sessions scheduled acording the study protocol
Number of scheduled visits attended | 6 months
  Number of visits attended by the patients out of the total of scheduled visits
Number of questionnaires fulfilled | 6 months
  Number of questionnaires fulfilled by the patients out of the total scheduled questionnaires
Number of telematics multidisciplinary sessions attended | 6 months
  Number of telematics multidisciplinary sessions attended by the patients out of the total scheduled sessions
Number of withdrawals | 6 months
  Number of withdrawals out of the total patients enrolled in the study

SECONDARY OUTCOMES:
SF-36 (Short Form-36) total punctuation | 6 months
  Quality of Life will be assessed by the SF-36 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Iago Garreta-Catala, MD, Principal Investigator — Orthopaedics Attending physician
Locations (1):
- Hospital de Bellvitge, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hurwitz EL, Randhawa K, Yu H, Cote P, Haldeman S. The Global Spine Care Initiative: a summary of the global burden of low back and neck pain studies. Eur Spine J. 2018 Sep;27(Suppl 6):796-801. doi: 10.1007/s00586-017-5432-9. Epub 2018 Feb 26. PMID 29480409
- [Result] Latremoliere A, Woolf CJ. Central sensitization: a generator of pain hypersensitivity by central neural plasticity. J Pain. 2009 Sep;10(9):895-926. doi: 10.1016/j.jpain.2009.06.012. PMID 19712899
- [Result] Searle A, Spink M, Ho A, Chuter V. Exercise interventions for the treatment of chronic low back pain: a systematic review and meta-analysis of randomised controlled trials. Clin Rehabil. 2015 Dec;29(12):1155-67. doi: 10.1177/0269215515570379. Epub 2015 Feb 13. PMID 25681408
- [Result] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Result] Meucci RD, Fassa AG, Faria NM. Prevalence of chronic low back pain: systematic review. Rev Saude Publica. 2015;49:1. doi: 10.1590/S0034-8910.2015049005874. Epub 2015 Oct 20. PMID 26487293
- [Result] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Derived] Garreta-Catala I, Planas-Balague R, Abouzari R, Carnaval T, Nolla JM, Videla S, Agullo-Ferre JL; EN-FORMA study group. Feasibility of a multidisciplinary group videoconferencing approach for chronic low back pain: a randomized, open-label, controlled, pilot clinical trial (EN-FORMA). BMC Musculoskelet Disord. 2023 Aug 9;24(1):642. doi: 10.1186/s12891-023-06763-6. PMID 37558990